CLINICAL TRIAL: NCT05782296
Title: Noninvasive Monitoring of Uterine Activity and Fetal Heart Rate: TrueLabor™, A New External Monitoring Device: Prospective Observational Study
Brief Title: Noninvasive Monitoring of Uterine Activity and Fetal Heart Rate
Status: Completed | Type: Observational
Sponsor: OB-Tools Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL-00002
Record Dates: First submitted 2022-02-28; First posted 2023-03-23 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Fetal Heart Rate or Rhythm Abnormality Affecting Newborn During Labor; Uterine Contractions; Obstetric Complication
Keywords: Fetal Heart Rate; Uterine Activity; TrueLabor; OB Tools; Non invasive monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Women in active labor following rupture of membranes and placement of an IUPC and/or FSE for obstetric indications
  Interventions: Device: TrueLabor

INTERVENTIONS:
Device: TrueLabor — Non invasive monitoring device

SUMMARY:
A clinical study designed to validate the safety and performance of the TrueLabor™ device in monitoring labor vs. current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Women who are on >=37w0d of gestation
* Maternal age > 18 years old
* Singleton pregnancy
* Cephalic presentation
* Patient requiring internal monitoring for obstetric indications
* Informed consent

Exclusion Criteria:

* Major fetal anomalies
* Patients with implanted electronic devices of any kind
* Patients using exterior electronic devices of any kind during the procedure
* Patients with irritated skin or open wound on the abdominal wall

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women in active labor
Study Population: Women (age>18 y/o) in active labor following rupture of membranes and placement of an IUPC and/or FSE.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Safety, comparative performance, and reliability of the TrueLabor™ system for Fetal Heart Rate | Through labor, until delivery
  This will be performed using a Performance Goal
Safety, comparative performance, and reliability of the TrueLabor™ system for Uterine Activity | Through labor, until delivery
  This will be performed using a Performance Goal

SECONDARY OUTCOMES:
Effect of BMI (weight in Kg, height in meters will be combined to report BMI in kg/m2) | Through labor, until delivery
  Effect of BMI on the performance measures

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Ascension Illinois Saint Alexius Residency Program in Obstetrics and Gynecology, Hoffman Estates, Illinois
  - Montefiore Medical Center, The Bronx, New York
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: OB Tools website — https://ob-tools.com/